CLINICAL TRIAL: NCT05244915
Title: Development and Feasibility of a Supportive Care Intervention for Older Caregivers of Older Adults with Advanced Cancer
Brief Title: A Supportive Care Intervention for Older Caregivers of Older Adults with Advanced Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been closed to accrual earlier than anticipated and will not resume.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Sindhuja Kadambi, Senior Instructor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS21067
Record Dates: First submitted 2021-08-03; First posted 2022-02-17 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-02

CONDITIONS: Cancer
Keywords: Cancer; Geriatric Assessment
MeSH Terms: conditions — Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Participants will receive a geriatric assessment which consists of validated questionnaires that are used to assess health status of older adults with cancer. Based on participant responses, tailored recommendations will be provided.
  Interventions: Other: Experimental (Delphi Surveys); Other: Experimental (Focus Groups); Other: Qualitative interviews

INTERVENTIONS:
Other: Experimental (Delphi Surveys) — The Delphi method, a process used to arrive at a group opinion or decision by surveying a panel of experts, will be used with experts in geriatric oncology to develop a supportive care management intervention for older caregivers of older adults with cancer.
Other: Experimental (Focus Groups) — Focus group qualitative interviews will be conducted with key stakeholders consisting of older adults with cancer and their caregivers.
Other: Qualitative interviews — Qualitative interviews will be conducted with older caregivers of older adults with cancer to inquire about their experience with caregiving and unmet supportive care needs.

SUMMARY:
This project assesses the feasibility of utilizing the geriatric assessment as a tool to identify distressed older caregivers of older adults with cancer. The investigator will engage key stakeholders including older caregivers of older adults with cancer, experts in geriatric oncology and primary care physicians to develop and pilot a supportive care intervention to improve outcomes in older caregivers.

DETAILED DESCRIPTION:
Older caregivers of older adults with cancer (described here-on as "older caregivers") are at high risk for increased burden and negative physical and psychological outcomes. Despite this, identification of older caregivers at risk for burden remains a challenge and evaluation of supportive care interventions and guidelines for this population remains limited. Health outcomes of older adults with cancer and their caregivers are inter-related and it is important to evaluate and support the health of both. The geriatric assessment (GA) is a valuable tool to evaluate health and age-related conditions (e.g., physical and cognitive function) of older adults with cancer and guide supportive care. Identifying older adults with age-related conditions can help to identify caregivers who are at increased risk for the negative impacts of caregiving. This project seeks to gather preliminary data on the health of older caregivers and to develop and pilot high priority supportive care interventions for this population. The investigator will examine the feasibility of utilizing the GA as a tool to identify distressed older caregivers. The investigator will engage key stakeholders including, older caregivers and older adults with cancer, experts in geriatric oncology and primary care physicians to develop and pilot a supportive care intervention to improve outcomes in older caregivers.

ELIGIBILITY:
Patient Inclusion Criteria

* Patient and caregiver be aged 65 or older
* Patient with a diagnosis of solid tumor malignancy or lymphoma, any stage
* Patients who have initiated a new line of treatment (surgery, radiation therapy, chemotherapy, immunotherapy, or targeted therapy) OR are being considered for new line of treatment (surgery, radiation therapy, chemotherapy, immunotherapy, or targeted therapy).
* Patients and caregivers must be able to provide informed consent, or if it is determined that they do not have decision-making capacity, a patient-designated health care proxy must sign consent per institutional University of Rochester and Research Subject Review Board policies on consent for incapacitated/decisionally impaired subjects.

Patient Exclusion Criteria

* Patient or caregiver is less than 65 years of age
* Patient and caregivers who do not have decision-making capacity (decisionally or cognitively impaired) AND do NOT have a previously designated health care proxy available to sign consent.

Caregiver Inclusion Criteria

* Caregivers enrolled in phase I
* Patient and caregiver have completed a GA

Caregiver Exclusion Criteria

• Patient and caregiver have not completed a GA

Stakeholder Inclusion Criteria

* Member of SCOREboard Community Advisory Board
* Aged 65 years or older
* Has been a family member, partner, friend or caregiver to an older adult with cancer

Stakeholder Exclusion Criteria • None

Geriatric Oncology Expert Inclusion Criteria

* Members of the Cancer and Aging Research Group
* Primary care physicians who care for older adults

Geriatric Oncology Expert Exclusion Criteria

• None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who enroll and complete the GA | 8 weeks per participant
  Percentage of participants who were approached, enrolled in the study and completed the GA will be determined.
Time for caregivers to complete the GA | 8 weeks per patient
  Time to complete the GA per caregiver will be determined by summing the time to complete self-administered and clinic portions of GA.
Caregiver satisfaction with completing the GA | 8 weeks per patient
  Caregivers will complete a questionnaire to assess satisfaction with completing the GA

SECONDARY OUTCOMES:
Percentage of caregiver supportive care recommendations that are implemented by patient/caregiver physicians | 4 weeks
  Caregivers will be surveyed to determined number and types of supportive care they received from their clinical providers compared to the supportive care recommendations that were provided to their clinical providers.

CONTACTS AND LOCATIONS:
Overall Officials: Sindhuja Kadambi, Principal Investigator — Univ. of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete and final study protocol will be made publicly available through the University of Rochester Cancer Center Community Oncology Research Program Research Base Protocol and Data Sharing Committee. The full protocol and data will be made publicly available no later than the publication date of the study findings from the final dataset. The protocol will include a detailed description of the study population, hypotheses tested, measurement and assessment information, data definitions and codes, and the analysis plan utilized. We will be collecting identifying information. The final dataset will be stripped of identifiers prior to release for sharing. Published papers will be made available in portable document format.
Time Frame: The data will be available for 7 years from accrual of the first subject.